CLINICAL TRIAL: NCT02578849
Title: Common Noradrenergic Mechanisms in Parkinson´s Disease and L-DOPA Induced Dyskinesia and Healthy Age Matched Controls; [11C]Yohimbine and [11C]MeNER PET
Brief Title: Common Noradrenergic Mechanisms in Parkinson´s Disease and L-DOPA Induced Dyskinesia
Acronym: NORAPARK
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aarhus University Hospital (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Adjmal Nahimi, MD, PhD, Aarhus University Hospital
Other Study IDs: 0602_Parkinson´s disease
Record Dates: First submitted 2015-09-30; First posted 2015-10-19 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-10

CONDITIONS: Parkinson´s Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Levodopa; carbidopa, levodopa drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- PD_no_LID: Patients with Parkinson´s disease without dyskinesia
  Interventions: Drug: L-DOPA
- PD_LID: Patients with Parkinson´s disease with L-DOPA induced dyskinesia
  Interventions: Drug: L-DOPA
- HC: Health controls, age-mathced.
  Interventions: Drug: L-DOPA

INTERVENTIONS:
Drug: L-DOPA — Patients and healthy controls are recruited to participate in [11C]yohimbine scans before and after L-DOPA challenge.
  Other Names: Sinemet

SUMMARY:
The aims of this proposal include tests of hypotheses of the pathogenetic mechanisms of noradrenergic neurotransmission in Parkinson's disease in vivo, using positron emission tomography of patients with early and advanced Parkinson's disease with or without 3,4 L-dihydroxyphenylalanine (L-DOPA) - induced dyskinesia or co-morbid depression, and evaluation of whether these mechanisms can be influenced therapeutically.

Hypotheses:

1. The investigators argue that release in human cortical and subcortical brain regions of norepinephrine (NE) derived from metabolism of exogenousL-DOPA is greater in Parkinson's disease patients with L-DOPA- induced dyskinesia than in patients without this complication. This hypothesis will be tested by measuring antagonist [11C]yohimbine binding to alpha-2 adrenoceptors before and after L-DOPA challenge.
2. If so, it is argued that the greater rise of norepinephrine, measured as [11C]yohimbine displacement after L-DOPA challenge, is the result of down-regulation or loss of norepinephrine transporters. This hypothesis will be tested by measuring the binding of [11C]MeNER, a tracer of norepinephrine transporters.
3. If so, the investigators argue that the greater decline of [11C]MeNER binding is significantly correlated to the symptoms of Parkinson's disease, as proof that patients with more severe loss of noradrenergic terminals exhibit more severe motor deficits.

DETAILED DESCRIPTION:
Introduction: The major source of NE in the central nervous system (CNS) is the locus coeruleus (LC), which sends projections to virtually all parts of the CNS, integrating cognitive and autonomic functions with the state of arousal (Sara SJ 2009).

With the onset of pathogenesis of PD in the lower brainstem, early symptoms of PD that include sleep disorder, cognitive deficits, and autonomic dysfunction, may appear prior to the motor symptoms of PD, and these symptoms have been linked to the degeneration of the LC and subsequent loss of noradrenergic innervations in the peripheral and central nervous systems (Rascol et al., 2009, Hawkes et al., 2010, Braak et al., 2003).

The loss of neurons in the LC exceeds that of the substantia nigra in some studies (Zarow et al. 2003), in which it is also argued that the loss may be related to the symptoms of endogenous depression in 40% of patients with PD. In these patients, the severity of motor symptoms also may be aggravated by loss of NE as release of dopamine (DA) and firing of dopaminergic neurons normally are both facilitated by activation of noradrenergic neurons.

Lesion of the LC and the subsequent loss of this facilitation reduces nigrostriatal DA release. Similarly, lesions to both dopaminergic and noradrenergic neurons induce more severe motor deficits, compared to lesions of dopaminergic neurons alone (Mavridis M et al., 1999). This relation suggests direct and indirect roles for NE in the emergence and severity of both motor and non-motor symptoms in PD, including depression.

The effects of NE are mediated by stimulation of the three receptor subtypes alpha-1, alpha-2, and ß. In the proposed studies, the investigators focus on alpha-2 and ß-receptors. Of the alpha-2 receptors, the alpha2C subtype is densely expressed in structures of the basal ganglia and therefore may mediate the direct effects of alpha-2 receptors on motor behavior.

However, in contrast to the possible beneficial effects of NE receptor activation in some brain regions, non-physiological increases of NE, after L- DOPA administration, may elicit dyskinesia (Buck et al., 2010) while fluctuations of NE concentration in other regions may contribute to generation of symptoms of depression (Zarow et al. 2003). Thus, several lines of evidence suggest that loss of NE may have direct and indirect roles in the appearance and severity of both motor and non-motor symptoms of PD and in LIDs.

Background:

Noradrenergic treatment of PD: The initial relief from symptoms of PD offered by DA agonist therapy is complicated by the manifestation of motor fluctuations, dyskinesia and psychiatric side effects following chronic treatment (Ahlskog et al., 2001, Fox et al., 2008).

The efficacy of conventional DA agonist therapy to reduce motor symptoms in PD is related to its ability to restore lost dopaminergic innervations. However, recent evidence suggests that activation of non- dopaminergic transmitter systems, including the noradrenergic system may play an important role in mediating the anti-parkinsonian effects of L-DOPA. L-DOPA and DA are sequential precursors of NE, and excitation of noradrenergic receptors following L-DOPA administration may contribute to the anti-parkinsonian effects of L-DOPA ( Schapira et al., 2008). Non-physiologically high release of NE derived from exogenous L-DOPA derived NE may contribute to both co-morbid depression and LID.

It further suggests that therapies that maintain L-DOPA- induced activation of NE receptors at physiological levels would reduce the severity of LID in patients. However, the underlying mechanisms of possible anti-parkinsonian and dyskinetogenic roles of NE remain unresolved. In this project, the investigators propose to identify the mechanisms through which NE conveys both beneficial and adverse effects of L-DOPA in a concerted attempt to help improve current treatment of PD by suggesting therapies that target the non-physiological L- DOPA-induced activation of the NE receptors as a potential contributor to LID.

The investigators developed and validated a novel PET tracer to be used in this project. Carbon-11 labelled yohimbine is an alpha-2 adrenoceptor antagonist and have been validated in studies with PET in pigs (Jakobsen et al., 2006, Landau et al. 2012) and approved for human use. To show that binding of [11C]yohimbine is sensitive to endogenously released NE, the investigators determined the binding before and after Vagus Nerve Stimulation in minipigs in vivo.

This group of researchers also developed the selective NET ligand, [11C]MeNER, for clinical PET studies in Denmark. Patients with PD and age-matched healthy controls will undergo PET-scans with the above-mentioned tracers to map pathological changes in noradrenergic transporters and receptors in-vivo.

ELIGIBILITY:
Inclusion Criteria:

* 15 patients with PD in the age between 50 og 80, Hoehn og Yahr stage 2-3, never L-DOPA induced dyskinesia.
* 15 patients with PD in the age between 50 og 80 år, Hoehn og Yahr stage 2-3, with established L-DOPA induced dyskinesia.
* 15 age matched healthy controls.

Exclusion Criteria:

* Psychiatric or neurological disease, not related to Parkinson´s disease.
* Cancer and malignant disease.
* Liver or kidney disease.
* Alcohol or substance abuse.
* Cardiac disease.
* Treatment with antipsychotics or antiepileptics or other medications that affect the noradrenergic system. Medicines to treat Parkinson´s disease are allowed.
* Patients treated with deep brain stimulation.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Parkinson´s disease patients with/without L-DOPA induced dyskinesia and age-matched healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2012-01; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Noradrenaline release | Up to 16 months
  Quantification of noradrenaline release in patients with Parkinson´s disease and healthy controls after pretreatment with 150mg L-DOPA as evaluated with [11C]yohimbine positron. emission tomography.

SECONDARY OUTCOMES:
Noradrenaline transporters | Up to 16 months
  Correlation of peripheral loss of noradrenaline in the heart with loss of central noradrenergic neurons in patients with Parkinson´s disease.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nuclear Medicine and PET-Centre, Aarhus University Hospital, Aarhus C, Denmark, Denmark

REFERENCES:
- [Result] Sara SJ. The locus coeruleus and noradrenergic modulation of cognition. Nat Rev Neurosci. 2009 Mar;10(3):211-23. doi: 10.1038/nrn2573. Epub 2009 Feb 4. PMID 19190638
- [Result] Rascol O, Schelosky L. 123I-metaiodobenzylguanidine scintigraphy in Parkinson's disease and related disorders. Mov Disord. 2009;24 Suppl 2:S732-41. doi: 10.1002/mds.22499. PMID 19877202
- [Result] Hawkes CH, Del Tredici K, Braak H. A timeline for Parkinson's disease. Parkinsonism Relat Disord. 2010 Feb;16(2):79-84. doi: 10.1016/j.parkreldis.2009.08.007. Epub 2009 Oct 28. PMID 19846332
- [Result] Braak H, Del Tredici K, Rub U, de Vos RA, Jansen Steur EN, Braak E. Staging of brain pathology related to sporadic Parkinson's disease. Neurobiol Aging. 2003 Mar-Apr;24(2):197-211. doi: 10.1016/s0197-4580(02)00065-9. PMID 12498954
- [Result] Buck K, Ferger B. Comparison of intrastriatal administration of noradrenaline and l-DOPA on dyskinetic movements: a bilateral reverse in vivo microdialysis study in 6-hydroxydopamine-lesioned rats. Neuroscience. 2009 Mar 3;159(1):16-20. doi: 10.1016/j.neuroscience.2008.12.026. Epub 2008 Dec 24. PMID 19146929
- [Result] Ahlskog JE, Muenter MD. Frequency of levodopa-related dyskinesias and motor fluctuations as estimated from the cumulative literature. Mov Disord. 2001 May;16(3):448-58. doi: 10.1002/mds.1090. PMID 11391738
- [Result] Fox SH, Lang AE, Brotchie JM. Translation of nondopaminergic treatments for levodopa-induced dyskinesia from MPTP-lesioned nonhuman primates to phase IIa clinical studies: keys to success and roads to failure. Mov Disord. 2006 Oct;21(10):1578-94. doi: 10.1002/mds.20936. PMID 16874752
- [Result] Schapira AH, Olanow CW. Drug selection and timing of initiation of treatment in early Parkinson's disease. Ann Neurol. 2008 Dec;64 Suppl 2:S47-55. doi: 10.1002/ana.21460. PMID 19127579
- [Result] Jakobsen S, Pedersen K, Smith DF, Jensen SB, Munk OL, Cumming P. Detection of alpha2-adrenergic receptors in brain of living pig with 11C-yohimbine. J Nucl Med. 2006 Dec;47(12):2008-15. PMID 17138744
- [Result] Landau AM, Dyve S, Jakobsen S, Alstrup AK, Gjedde A, Doudet DJ. Acute Vagal Nerve Stimulation Lowers alpha2 Adrenoceptor Availability: Possible Mechanism of Therapeutic Action. Brain Stimul. 2015 Jul-Aug;8(4):702-7. doi: 10.1016/j.brs.2015.02.003. Epub 2015 Feb 13. PMID 25758422